CLINICAL TRIAL: NCT07366931
Title: A Randomized, Placebo-controlled, Double-blind Trial on the Effect of Daily Supplementation With Humiome® Post LB on Gastrointestinal Symptoms in Female Athletes
Brief Title: The Effect of Daily Supplementation With Humiome® Post LB on Gastrointestinal Symptoms in Female Athletes
Acronym: GI-Jane
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Kat Silang, Research Assistant, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25/SPS/057
Record Dates: First submitted 2025-12-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Females; Gastrointestinal Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator)
  Interventions: Drug: Postbiotic
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Postbiotic — Participants allocated to this arm will receive the investigational product (Humiome(R) Post LB), to be ingested daily for three consecutive menstrual cycles.
  Arms: Active
Drug: Placebo — Participants allocated to this arm will receive a visually identical placebo to the verum, to be ingested daily for three consecutive menstrual cycles.
  Arms: Placebo

SUMMARY:
Female athletes are often overlooked in scientific research, including the understanding of their digestive system and its impact on overall health, training, and performance. The gastrointestinal (GI) system plays a critical role in supporting digestion, nutrient absorption, and acting as a protective barrier for the body. While there is some knowledge about the differences in GI structure and function between males and females at rest, there is a lack of understanding regarding how these differences manifest during exercise, especially among female athletes and at different phases of the menstrual cycle.

It has been observed that female athletes commonly report a higher prevalence of GI symptoms compared to males, with many experiencing an increase during menstruation. These symptoms, including bloating, abdominal discomfort, and irregular bowel movements, can significantly disrupt an athlete's training and performance. Elite female athletes have acknowledged that GI symptoms associated with the menstrual cycle have led to altered or disrupted training routines. While these symptoms are commonly recognized to affect a large portion of the female population, few interventions have been studied to assist in managing this discomfort. Some clinicians may direct their patients to take pain-relieving medications without any thoughts on the consequences of chronic use.

One potential strategy to reduce GI symptoms during endurance exercise is probiotic-postbiotic supplementation. Various probiotic supplements have been shown to effectively decrease diarrhoea, constipation stress, and intestinal permeability, as well as impact immunologic outcomes. Postbiotics differ from probiotics in that they are made from microorganisms that are not alive. They allow the modulation of the composition and function of the gut microbiota and enhance the intestinal barrier to prevent unwanted substances from entering the body proper. While these biotics can relieve lower GI symptoms in irritable bowel syndrome (IBS), there is less consensus regarding their efficacy in modulating exercise-associated GI symptoms. Previous research by Pugh et al., 2019 has demonstrated that four weeks of probiotic supplementation was able to reduce GI symptoms during a marathon race, however this work was predominantly conducted in males and did not take menstrual cycle in consideration. This is important given that symptoms are commonly higher in the early follicular phase when a female experiences their period. Therefore, the aim of this study is to assess the effects of postbiotic supplementation on GI symptomology in female athletes.

The aim of this present study is to investigate the influence of postbiotic supplementation on menstrual cycle symptoms and exercise-associated GI symptoms in female endurance athletes while exercising compared to symptoms while taking a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Female, cisgender, premenopausal.
2. Minimum age 18 years.
3. Regular, natural menstrual cycle (21-35 days in duration), with 9 or more consecutive periods per year, if possible documented with tracker apps, calendars, or other tools.
4. Willingness and ability to give informed consent and to understand, to participate, and to comply with the clinical study requirements.
5. Body mass index (BMI) ≥ 18.5 and < 24.9 kg/m2
6. Agreeing to maintain lifestyle habits during the study (same dietary and physical activity habits)
7. Having a smartphone and a history of consistent tracking of training and health records via apps.
8. Having regular GI issues during exercise, preferably also during menstruation. During pre-screening, this will be assessed with a shortened GSRS questionnaire, where participants need to have had, in the month preceding pre-screening, the equivalent of at least a score of 2 in a GSRS focus area (diarrhoea, pain, indigestion).
9. No relevant self-reported abnormalities from medical history.
10. Trained athlete (trains at least 3 times per week for more than 1 hour per day and who has been involved in endurance training for at least 2 years in alignment with previous research (Pfeiffer et al., 2010). This will be evaluated by assessing training records (Strava or similar application, certificates of attendance to athletic events, club membership, etc.).
11. Access to a health-care provider, who can be contacted by the CRO, and who reside in areas with available health services.

Exclusion Criteria:

1. Individuals who are pregnant, lactating, or plan to become pregnant before study end.
2. Individuals with secondary amenorrhea.
3. Individuals who use hormonal contraceptives during the last 6 months before (and during) the trial.
4. Individuals who are currently participating in another clinical trial or have participated in a trial within the last two months prior to enrolment.
5. Tobacco smokers and vapers.
6. Individuals with acute illness.
7. Individuals with a current musculoskeletal injury or one within the last month.
8. Individuals taking probiotic supplements or who have taken probiotics two weeks prior to enrolment.
9. Individuals controlling chronic diseases with treatments known to alter the intestinal microbiome or to alter GI symptoms, such as certain pain killers, antacids, proton-pump inhibitors, anti-diarrhoeal medication or supplements, and laxatives.
10. Individuals having received antibiotics treatments within three months of trial start.
11. Individuals having planned major changes in lifestyle (i.e. diet, weight loss program, exercise level, travelling) during the duration of the study.
12. Individuals who have any hypersensitivity/allergy to any of the components of the test product.
13. Individuals who have planned major elective surgery during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS) scores | Starting from Day 1 of the participants' menstrual cycle, the questionnaire is to be completed every seven days for the duration of the trial, an average of three months.
  A list of fifteen gastrointestinal symptoms scored on a Likert scale, where 1=no discomfort at all, and 7=very severe discomfort.

SECONDARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS) Sub-scores | Starting from Day 1 of the participants' menstrual cycle, the questionnaire is to be completed every seven days for the duration of the trial, an average of three months.
  A list of fifteen gastrointestinal symptoms scored on a Likert scale, where 1=no discomfort at all, and 7=very severe discomfort. The symptoms are grouped into five sub-categories: Reflux, Abdominal pain, Indigestion, Diarrhoea, and Constipation.
Wilson Gastrointestinal (GI) Score | Questionnaire to be completed once a day on the days the participants are menstruating. An average of 5 days every cycle, for the duration of the trial, an average of three months.
  A list of six gastrointestinal symptoms scored on a Likert scale, with the following descriptors:
  0=no discomfort 5=moderate discomfort 10=unbearable discomfort.
Faecal microbiome composition | Two times throughout participation (average of three months); first sample is taken after the first month of participation, and second sample taken after the third month of participation. Exact times vary from participant to participant.
  Faecal samples will be collected to assess gut microbial composition using full shotgun sequencing.
Faecal microbiome diversity | Two times throughout participation (average of three months); first sample is taken after the first month of participation, and second sample taken after the third month of participation. Exact times vary from participant to participant.
  Faecal samples will be collected to assess gut microbial diversity using full shotgun sequencing.
Adherence to physical activity training schedules | Starting from Day 1 of the participants' menstrual cycle, the diary is to be completed every seven days for the duration of the trial, an average of three months.
  Participants will be asked to complete a weekly training diary where they will provide any planned training activities and their adherence to these plans. Data taken will be minutes of activity per week and intensity of the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pugh JN, Sparks AS, Doran DA, Fleming SC, Langan-Evans C, Kirk B, Fearn R, Morton JP, Close GL. Four weeks of probiotic supplementation reduces GI symptoms during a marathon race. Eur J Appl Physiol. 2019 Jul;119(7):1491-1501. doi: 10.1007/s00421-019-04136-3. Epub 2019 Apr 13. PMID 30982100
- [Background] Pugh JN, Lydon KM, O'Donovan CM, O'Sullivan O, Madigan SM. More than a gut feeling: What is the role of the gastrointestinal tract in female athlete health? Eur J Sport Sci. 2022 May;22(5):755-764. doi: 10.1080/17461391.2021.1921853. Epub 2021 May 20. PMID 33944684
- [Background] Judkins TC, Dennis-Wall JC, Sims SM, Colee J, Langkamp-Henken B. Stool frequency and form and gastrointestinal symptoms differ by day of the menstrual cycle in healthy adult women taking oral contraceptives: a prospective observational study. BMC Womens Health. 2020 Jun 29;20(1):136. doi: 10.1186/s12905-020-01000-x. PMID 32600463
- [Background] Hungin APS, Mitchell CR, Whorwell P, Mulligan C, Cole O, Agreus L, Fracasso P, Lionis C, Mendive J, Philippart de Foy JM, Seifert B, Wensaas KA, Winchester C, de Wit N; European Society for Primary Care Gastroenterology. Systematic review: probiotics in the management of lower gastrointestinal symptoms - an updated evidence-based international consensus. Aliment Pharmacol Ther. 2018 Apr;47(8):1054-1070. doi: 10.1111/apt.14539. Epub 2018 Feb 20. PMID 29460487
- [Background] Bruinvels G, Goldsmith E, Blagrove R, Simpkin A, Lewis N, Morton K, Suppiah A, Rogers JP, Ackerman KE, Newell J, Pedlar C. Prevalence and frequency of menstrual cycle symptoms are associated with availability to train and compete: a study of 6812 exercising women recruited using the Strava exercise app. Br J Sports Med. 2021 Apr;55(8):438-443. doi: 10.1136/bjsports-2020-102792. Epub 2020 Nov 16. PMID 33199360
- [Background] Brown N, Knight CJ, Forrest Nee Whyte LJ. Elite female athletes' experiences and perceptions of the menstrual cycle on training and sport performance. Scand J Med Sci Sports. 2021 Jan;31(1):52-69. doi: 10.1111/sms.13818. Epub 2020 Sep 19. PMID 32881097